CLINICAL TRIAL: NCT07190183
Title: Washed Microbiota Transplantation for Food Intolerance
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professsor, Gastroenterology, The Second Hospital of Nanjing Medical University
Other Study IDs: WMT-FI
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-01

CONDITIONS: Food Intolerance
Keywords: washed microbiota transplantation; food intolerance; fecal microbiota transplantation; gut microbiota
MeSH Terms: conditions — Food Intolerance | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — faeces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The FI undergoing washed microbiota transplantation: patients undergoing washed microbiota transplantation who were diagnosed as food intolerance according to laboratory examination
  Interventions: Procedure: washed microbiota transplantation
- The FI not undergoing washed microbiota transplantation: The FI did not undergo washed microbiota transplantation

INTERVENTIONS:
Procedure: washed microbiota transplantation — The prepared microbiota suspension was infused into the patients' gut.
  Other Names: fecal microbiota transplantation
  Groups: The FI undergoing washed microbiota transplantation

SUMMARY:
Food intolerance (FI) is an adverse reaction to food caused by non-immune mechanisms, mainly related to digestive enzyme deficiencies (e.g. lactase deficiency), metabolic abnormalities (e.g. impaired absorption of fructose) or toxicity of food components (e.g. histamine). Unlike immune-mediated food allergy, FI symptoms are usually delayed (hours to days after ingestion) and mild, but are difficult to diagnose and manage clinically due to the complexity and variety of mechanisms that affect approximately 20% of the world's population.

DETAILED DESCRIPTION:
The gut microbiota of food intolerance (FI) is different. The widespread use of artificial sweeteners (e.g. saccharin) can induce metabolic disorders by altering the structure of the intestinal flora, e.g. animal experiments have shown that the abundance of pathogenic bacteria (e.g. Bacteroides vulgatus) in the intestinal tract of mice ingesting saccharin was significantly increased, whereas the abundance of Akkermansia muciniphila was decreased, which led to impaired glucose tolerance and abnormal fat absorption, and ultimately increased the risk of obesity and diabetes mellitus. ultimately increasing the risk of obesity and diabetes . In addition, sorbitol, as a low-calorie sugar alcohol, can trigger osmotic diarrhoea when ingested in excess, while antibiotics combined with a high-fat diet further disrupts intestinal flora balance (e.g., Clostridia depletion), decreases flora sorbitol dehydrogenase activity, and leads to persistent sorbitol metabolism disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Food intolerance occurs through laboratory examination of at least two main foods
2. Underwent washed microbiota transplantation.

Exclusion Criteria:

1. Expected survival time <3 months;
2. Women who are pregnant or breastfeeding;
3. Other patients deemed not suitable for enrollment by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with food intolerance receiving WMT will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2035-02-10 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
change of weight and height | baseline, 4 weeks, 12 weeks post transplantation
  Weight and height will be combined to report BMI in kg/m^2.
change of the Gastrointestinal Symptom Rating Scale(GSRS) | baseline, 4 weeks, 12 weeks post transplantation
  GSRS is a 13-item test to make a comprehensive assessment of common gastrointestinal symptom and each item receives a value from 0 to 3, with higher value indicating worse gastrointestinal condition.

SECONDARY OUTCOMES:
change of insulin-like growth factor I(IGF-I),intestinal barrier function and immunoglobulin | baseline, 12 weeks post transplantation
  Blood test
the difference of the gut microbiota composition before and after washed microbiota transplantation | baseline, 12 weeks post transplantation
  The composition of the gut microbiota is evaluated by sequencing faecal metagenome. We evaluate the differences in the structure of the flora and its metabolism.
the incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | 12 weeks post transplantation
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No